CLINICAL TRIAL: NCT01227538
Title: Towards Simple and Non-invasive Assessment of Residual Beta-cell Function in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Danijela Tatovic, Consultant in Diabetes and Endocrinology, University Hospitals Bristol and Weston NHS Foundation Trust
Other Study IDs: ME/2010/3452; 10/H0505/87 (Other: Berkshire REC)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes
Keywords: Beta cell reserve, urinary C peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stimulated urinary C peptide: Study will be designed to assess stimulated urinary C-peptide in comparison to mixed-meal stimulated plasma C-peptide response in the same individual in 30 number of patients with Type 1 diabetes.
  Interventions: Other: Mixed meal stimulated urinary C peptide for the assessment of residual beta cell function

INTERVENTIONS:
Other: Mixed meal stimulated urinary C peptide for the assessment of residual beta cell function — Study will be designed to assess stimulated urinary C-peptide in comparison to mixed-meal stimulated plasma C-peptide response in the same individual in 30 number of patients with Type 1 diabetes.

SUMMARY:
Type 1 diabetes is condition in which progressive autoimmune destruction of insulin-producing beta-cells leads to absolute insulin deficiency. At the time of clinical presentation, it is estimated that 50-80% of beta-cell function has been lost. Good glycaemic control from diagnosis has been shown to preserve beta-cell function. The recent identification of immuno-interventions able to reduce autoimmune destruction and preserve beta-cell function has lead to an increased urgency to develop such tools.

With mixed-meal stimulated serum C-peptide being a gold standard, there are currently no tests that are suited for use in clinical practice to detect and monitor residual beta cell function. There is a therefore a need for a test that is sufficiently sensitive to assess beta cell function reserve in Type 1 diabetes for clinical practice purposes, which will be simple, reproducible and suitable for use even in the non-observed setting.

Using mixed meal stimulation of plasma C-peptide (stable by-product in insulin secretion that reliably reflects insulin production) response as a reference, we propose to compare mixed meal stimulated urinary C-peptide as potential candidate for this application. This is a pilot investigation in which a sample of 30 participants will be recruited.

It is anticipated that the current project will identify a simple method for analysing beta cell reserve in Type 1 diabetes. This will then be applied to screening clinic populations of recently diagnosed patients with type 1 diabetes. The aim will be to identify subjects who may be suitable for early intensified insulin regimes (e.g. insulin pump therapy) and novel immuno-intervention strategies designed to preserve residual beta cell function and improve long-term outcomes. Currently such immunointervention has been reserved for subjects within 3 months of diagnosis only, excluding a significant number of subjects who may potentially benefit.

ELIGIBILITY:
Inclusion Criteria:1. 1. Type 1 diabetes diagnosed in the last 5 years 2. Age 18-45 years 3. BMI between 18.5 and 29.9 4. Insulin requirement less than 0.8 units/kg

-

Exclusion Criteria:

1. HbA1c higher than 10% 2. Ongoing steroid treatment or chemotherapy 3. Pregnancy and breast feeding 4. eGFR less than 50ml/min/1.73m2

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with Type 1 diabetes diagnosed in the last 5 years
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of whether two-hour urinary C-peptide response to mixed-meal (measured as area under the curve on the graph) can be used assess residual beta-cell function in the first 5 years after diagnosis of Type 1 diabetes. | One year

SECONDARY OUTCOMES:
To compare fasting urinary C-peptide to plasma C-peptide response to mixed-meal | One year
To compare urinary C-peptide response to mixed meal in each hour post stimulation to plasma C-peptide response to mixed-meal | One year
To compare total four-hour urinary C-peptide (area under the curve) response to mixed meal to plasma C-peptide response to mixed-meal | One year
To assess whether urinary C-peptide response to mixed-meal is reproducible in non-observed setting. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Clinical Research Unit, UHBristol NHS Foundation Trust, Bristol, Avon, United Kingdom